CLINICAL TRIAL: NCT03125629
Title: Comparison of PET/CT vs. PET/MRI
Brief Title: Comparison of PET/CT vs. PET/MRI Using 2 Radiopharmaceuticals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrei Iagaru, Associate Professor of Radiology, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-27398; NCI-2017-00364 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VARIMG0004 (Other: OnCore)
Record Dates: First submitted 2017-03-24; First posted 2017-04-24 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Cancer Diagnosis; Diagnostic Techniques and Procedures; Diagnostic Imaging
MeSH Terms: interventions — gallium Ga 68 dotatate; Positron-Emission Tomography; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography; Radionuclide Imaging; Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: All participants receive both scans.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- 18F-FDG PET/CT Scan (Experimental): Participants will undergo a PET/CT scan with radiolabel 18F-FDG.
  Interventions: Drug: F-18 FDG; Device: Positron Emission Tomography / Computed Tomography (PET/CT) Scan
- 18F-FDG PET/MRI Scan (Experimental): Participants will undergo a PET/MRI scan with radiolabel 18F-FDG.
  Interventions: Drug: F-18 FDG; Device: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) Scan
- 68Ga-DOTA-TATE PET/CT Scan (Experimental): Participants will undergo a PET/CT scan with radiolabel 68Ga-DOTA-TATE.
  Interventions: Drug: Ga-68-DOTA-TATE; Device: Positron Emission Tomography / Computed Tomography (PET/CT) Scan
- 68Ga-DOTA-TATE PET/MRI Scan (Experimental): Participants will undergo a PET/MRI scan with radiolabel 68Ga-DOTA-TATE.
  Interventions: Drug: Ga-68-DOTA-TATE; Device: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) Scan

INTERVENTIONS:
Drug: F-18 FDG — Radiolabel for positron emission tomography / computed tomography (PET/CT) and computed tomography (PET/CT) imaging
  Arms: 18F-FDG PET/CT Scan; 18F-FDG PET/MRI Scan
Drug: Ga-68-DOTA-TATE — Radiolabel for positron emission tomography / computed tomography (PET/CT) and computed tomography (PET/CT) imaging
  Arms: 68Ga-DOTA-TATE PET/CT Scan; 68Ga-DOTA-TATE PET/MRI Scan
Device: Positron Emission Tomography / Computed Tomography (PET/CT) Scan — Scan using a regular medical care (IDE-exempt) Discovery 600 / 690 PET/CT scanner.
  Arms: 18F-FDG PET/CT Scan; 68Ga-DOTA-TATE PET/CT Scan
Device: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) Scan — Scan using a NOVEL GE PET/MRI scanner.
  Arms: 18F-FDG PET/MRI Scan; 68Ga-DOTA-TATE PET/MRI Scan

SUMMARY:
This clinical trial studies how well positron emission tomography (PET)/computed tomography (CT) works compared to PET/magnetic resonance imaging (MRI) in evaluating patients with cancer. PET/CT and PET/MRI may determine which scanner is best for the patient's type of cancer and other types of cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if PET/CT and PET/MRI scanners provide equivalent results for evaluation of cancer patients.

OUTLINE:

Patients receive standard of care 18F-fludeoxyglucose (FDG) or Ga68-DOTA-TATE intravenously (IV). Within 45-60 minutes, patients then undergo PET/CT imaging immediately followed by PET/MRI. Each participant is to receive 18-FDG or 68Ga-DOTA-TATE only, no participant was to receive both radiotracers.

ELIGIBILITY:
INCLUSION CRITERIA

* Cancer diagnosis
* Capable of complying with study procedures
* Able to remain still for duration of imaging procedure (approximately 90 minutes total)
* Written informed consent

EXCLUSION CRITERIA

* Pregnant or nursing
* Metallic implants
* Impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-05-27 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2020-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Most subjects participated in more than 1 treatment arm. In order to not have participants represented multiple times in Participant Flow, this information is provided only at the study level.
Groups:
- Total Participant Flow: Participant Flow reflects participation of individual human participants. Individual participants are present in multiple assessment groups ("arms" or "cohorts").
Period: Overall Study
Arm/Group | Total Participant Flow
Started | 53
Completed | 50
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Equipment malfunction | 1

BASELINE CHARACTERISTICS:
Population: Most subjects participated in more than 1 treatment arm. In order to not have participants represented multiple times in Participant Flow, this information is provided only at the study level.
Groups:
- Total Participants: Baseline information reflects participation of the individual human participants. Individual human participants are present in multiple assessment groups ("arms" or "cohorts"), and to avoid over-representation of those participants, data is not reported by group.
Arm/Group | Total Participants
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.34 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Absolute Accuracy of SUV Max of PET/CT vs PET/MRI
Description: Standardized uptake value max (SUVmax) is a measurement of the maximum radiopharmaceutical uptake value within the region of interest (ROI). SUVmax is calculated as the ratio of activity concentration:injected dose/body weight. The outcome is reported as the mean SUVmax with standard deviation (SD), reported for 8 specific organs or bodily locations.
Time Frame: 4 hours
Population: Not all scans at all body locations could be completed.
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: scans
Arm/Group | 18F-FDG PET/CT Scan | 18F-FDG PET/MRI Scan | 68Ga-DOTA-TATE PET/CT Scan | 68Ga-DOTA-TATE PET/MRI Scan
Number analyzed (Participants) | 44 | 42 | 6 | 6
Number analyzed (scans) | 44 | 42 | 6 | 6
ratio
  Aortic arch: number analyzed (Participants) | 44 | 40 | 6 | 6
  Aortic arch: number analyzed (scans) | 44 | 40 | 6 | 6
  Aortic arch | 1.78 (0.42) | 1.08 (0.38) | 0.54 (0.22) | 0.51 (0.19)
  Gluteal muscle: number analyzed (Participants) | 44 | 41 | 6 | 6
  Gluteal muscle: number analyzed (scans) | 44 | 41 | 6 | 6
  Gluteal muscle | 0.79 (0.20) | 0.94 (0.28) | 0.42 (0.19) | 0.47 (0.25)
  Gluteal fat: number analyzed (Participants) | 44 | 41 | 6 | 6
  Gluteal fat: number analyzed (scans) | 44 | 41 | 6 | 6
  Gluteal fat | 0.27 (0.10) | 0.26 (0.09) | 0.14 (0.06) | 0.24 (0.07)
  Cerebellum: number analyzed (Participants) | 40 | 41 | 4 | 4
  Cerebellum: number analyzed (scans) | 40 | 41 | 4 | 4
  Cerebellum | 8.56 (2.64) | 7.79 (2.49) | 0.22 (0.09) | 0.12 (0.12)
  Parotid Gland: number analyzed (Participants) | 41 | 42 | 5 | 5
  Parotid Gland: number analyzed (scans) | 41 | 42 | 5 | 5
  Parotid Gland | 1.71 (0.68) | 1.76 (0.77) | 1.28 (0.60) | 1.06 (0.26)
  Lung | 0.57 (0.21) | 0.36 (0.15) | 0.31 (0.05) | 0.26 (0.20)
  Liver: number analyzed (Participants) | 44 | 41 | 6 | 6
  Liver: number analyzed (scans) | 44 | 41 | 6 | 6
  Liver | 2.72 (0.66) | 2.21 (0.59) | 9.47 (7.15) | 10.86 (7.60)
  Spleen: number analyzed (Participants) | 40 | 37 | 2 | 2
  Spleen: number analyzed (scans) | 40 | 37 | 2 | 2
  Spleen | 2.18 (0.82) | 2.03 (0.97) | 13.07 (3.75) | 15.74 (3.16)

2. Secondary Outcome: PET/CT vs PET/MRI Difference in Standardized Uptake Value Max (SUVmax), by Radiotracer
Description: Standardized uptake value max (SUVmax) is a measurement of the maximum radiopharmaceutical uptake within the region of interest (ROI). Relative accuracy of a particular radiotracer in a particular tissue is determined by expressing the absolute accuracy (obtained in the primary outcome measure) in terms of percent difference between SUVmax values obtained from PET/CT and PET/MR.
  Percentage difference is expressed as the difference of the means in SUVmax for the PET/CT and PET/MRI scan procedures for the particular radiotracer, divided by the mean between the values for the 2 scan procedures.
  The closer the percent difference is to 0%, the better the agreement between the two scanners. The outcome is expressed as the percentage difference, a number without dispersion.
Time Frame: estimated average of 2 hours
Population: Not all scans at all body locations could be completed.
Measure: Number; unit: Percentage difference
Units Other Than Participants: Scans (PET/CT + PET/MRI)
Groups:
- 18-FDG PET/CT and PET/MRI: PET/CT and PET/MRI scans were conducted using radiotracer 18-FDG.
- 68Ga DOTA-TATE PET/CT and PET/MRI: PET/CT and PET/MRI scans were conducted using radiotracer 68Ga DOTA-TATE.
Arm/Group | 18-FDG PET/CT and PET/MRI | 68Ga DOTA-TATE PET/CT and PET/MRI
Number analyzed (Participants) | 44 | 6
Number analyzed (Scans (PET/CT + PET/MRI)) | 86 | 12
Percentage difference
  Aortic arch: number analyzed (Scans (PET/CT + PET/MRI)) | 84 | 12
  Aortic arch | 48.95 | 5.71
  Gluteal muscle: number analyzed (Scans (PET/CT + PET/MRI)) | 85 | 12
  Gluteal muscle | 17.34 | 11.24
  Gluteal fat: number analyzed (Scans (PET/CT + PET/MRI)) | 85 | 12
  Gluteal fat | 3.77 | 52.63
  Cerebellum: number analyzed (Participants) | 41 | 4
  Cerebellum: number analyzed (Scans (PET/CT + PET/MRI)) | 81 | 8
  Cerebellum | 9.42 | 58.82
  Parotid Gland: number analyzed (Participants) | 42 | 5
  Parotid Gland: number analyzed (Scans (PET/CT + PET/MRI)) | 83 | 10
  Parotid Gland | 2.88 | 18.80
  Lung | 45.16 | 17.54
  Liver: number analyzed (Scans (PET/CT + PET/MRI)) | 85 | 12
  Liver | 20.69 | 13.67
  Spleen: number analyzed (Participants) | 40 | 2
  Spleen: number analyzed (Scans (PET/CT + PET/MRI)) | 77 | 4
  Spleen | 7.13 | 18.54

ADVERSE EVENTS:
Time Frame: 1 day
Description: Per protocol, only unanticipated adverse events were to be collected.
Arm/Group | 18F-FDG PET/CT Scan | 18F-FDG PET/MRI Scan | 68Ga-DOTA-TATE PET/CT Scan | 68Ga-DOTA-TATE PET/MRI Scan
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/42 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/44 | 0/42 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03125629/Prot_SAP_000.pdf